CLINICAL TRIAL: NCT04866966
Title: Shared Medical Appointments for Weight Loss
Acronym: SMALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: American College of Clinical Pharmacy (Other)
Responsible Party: Principal Investigator, Rachel B. Franks, Assistant Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00033354
Record Dates: First submitted 2018-12-03; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Shared Medical Appointments; Small-Area Analysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The group undergoing the intervention will participate in 90-minute group visits occurring weekly for 4 weeks, then biweekly for a total of 26 weeks/15 visits. Each visit will focus on intensive lifestyle changes. Further, these patients will each have the opportunity to meet one-on-one with a member of the research team at the end of each visit in order to discuss individual goals and progress. Pharmacotherapy therapy changes will be recommended to reduce or avoid use of medication which may contribute to weight gain and medications for weight loss will be prescribed as an individualized treatment strategy during one-on-one time with the pharmacist or physician if the patient can afford it and no contraindications exists.
  Interventions: Behavioral: Shared medical appointments for weight loss
- Control Group (No Intervention): The control group will have their measurements done at the beginning and end of the study. They will continue with usual medicare care during the study and will not receive any education from the investigators during the study. They will be offered the option of a delayed intervention after the completion of the study.

INTERVENTIONS:
Behavioral: Shared medical appointments for weight loss — Shared medical appointments providing education and lifestyle change recommendations to promote weight loss in obese patients
  Other Names: SMALL Study
  Arms: Intervention Group

SUMMARY:
Randomized controlled trial to determine if a 6 months of shared medical appointments will results in clinically and statistically significant weight loss.

DETAILED DESCRIPTION:
Obese patients will be randomized to either the control or intervention group. The intervention group will participate in 90-minute group visits occurring weekly for 4 weeks, then biweekly for a total of 26 weeks/15 visits. Each visit will focus on intensive lifestyle changes: calorie restriction to produce a 500-750 calorie deficit, increased physical activity, and behavioral therapies including regular self-monitoring of food intake, physical activity, and weight. Additional behavioral therapies that will be offered include techniques for reducing stress, maximizing sleep, and controlling environments. Further, these patients will each have the opportunity to meet one-on-one with a member of the research team at the end of each visit in order to discuss individual goals and progress.

ELIGIBILITY:
Inclusion Criteria:

* Current patients of the USF Family or General Internal Medicine Clinics
* BMI of 30 or greater
* Able to speak and read English

Exclusion Criteria:

* Age over 75 years, patients with end-stage renal disease with estimated GFR less than 15 mL/min, diabetes mellitus with an A1C > 9%, Acute Coronary Syndrome (such as unstable angina, pacemaker or defibrillator due to impedance scale), recent history of weight loss (>5% of body weight), pregnant or breastfeeding women, dementia or unstable psychiatric disorder, participation in any structured weight loss program currently or in the previous 3 months, cancer, or anyone unable to complete study protocol (exercise amounts, food intake).

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Percentage of participants from each group who lost at least 5% of their initial body weight | 6 months
  Body weight will be measured at the initial and final visits using the Tanita DC-430 body composition analyzer for participants in both groups and documented in the medical record. Percent of body weight lost will be calculated for each participant and the percentage of participants who lose 5% of body weight will be included in the primary outcome.

SECONDARY OUTCOMES:
Mean change in body weight from each group from baseline to the final visit | 6 months
  Body weight will be measured at the initial and final visits using the Tanita DC-430 body composition analyzer for participants in both groups and documented in the medical record. Change in weight will be calculated for each participant and the mean will be reported.
Mean percent weight change of each group from baseline to the final visit | 6 months
  Body weight will be measure at the initial and final visits using the Tanita DC-430 body composition analyzer for participants in both groups and documented in the medical record. Percent of body weight lost will be calculated for each participant and the mean will be reported.
Mean change in body mass index (BMI) of each group from baseline to the final visit | 6 months
  BMI will be calculated using weight and height measured at the initial and final visits and the difference will be calculated for each participant and documented in the medical record. Weights will be measured using the Tanita DC-430 body composition analyzer and heights measured using a stadiometer on a physicians scale. The mean for each group will be reported.
Mean change in body fat percentage of each group from baseline to final visit | 6 months
  The Tanita DC-430 body composition analyzer will be used to measure body fat percentages for each participant at the initial and final visits and documented in the medical record. The change will be calculated for each participant and the mean for each group will be reported.
Mean percentage of participants from each group without weight gain | 6 months
  Body weight will be measured at the initial and final visits using the Tanita DC-430 body composition analyzer for participants in both groups and documented in the medical record. The percentage of participants in each group who lost or does not gain weight during the study will be reported for each group.
Mean change in doses or number of medications for hypertension or diabetes | 6 months
  Weight loss or weight gain can affect the need for medications for diabetes and hypertension. The number and doses of medications for hypertension and type 2 diabetes will recorded in the medical record at the initial and final visits. The changes in number or dosage will be reported for each group.
Effect of visit adherence on each outcome | 6 months
  We will assess if or how visit attendance affects the results of each outcome per group. Attendance will be recording in the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel B Franks, PharmD, Principal Investigator — University of South Florida Health
Locations (1):
- Byrd Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No